CLINICAL TRIAL: NCT06685081
Title: Optimal-dose of Dexmedetomidine as Adjuvant to Epidural Local Anesthetic/Steroid Injectate to Improve Pain and Quality of Waking in Patients With Chronic Low Back Pain: A Randomized Case-control Study
Brief Title: Dexmedetomidine for Improved Pain Relief and Recovery in Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ahmed M Helwa, Lecturer of Anesthesia, Pain & ICU, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7-2024ANST5
Record Dates: First submitted 2024-11-11; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Lidocaine; Triamcinolone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group I (Active Comparator)
  Interventions: Drug: lidocaine and triamcinolone
- Group II (Active Comparator)
  Interventions: Drug: Dexmedetomidine; Drug: lidocaine and triamcinolone
- Group III (Active Comparator)
  Interventions: Drug: Dexmedetomidine; Drug: lidocaine and triamcinolone
- Group IV (Active Comparator)
  Interventions: Drug: Dexmedetomidine; Drug: lidocaine and triamcinolone
- Group V (Active Comparator)
  Interventions: Drug: Dexmedetomidine; Drug: lidocaine and triamcinolone

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine was injected in dose of 0.25 µg/kg
  Arms: Group II
Drug: Dexmedetomidine — Dexmedetomidine was injected in dose of 0.5 µg/kg
  Arms: Group III
Drug: Dexmedetomidine — Dexmedetomidine was injected in dose of 0.75 µg/kg
  Arms: Group IV
Drug: Dexmedetomidine — Dexmedetomidine was injected in dose of 1 µg/kg
  Arms: Group V
Drug: lidocaine and triamcinolone — 2 ml of 1.5% lidocaine and 2 ml of triamcinolone was mixed and provided to all patients as epidural injection

SUMMARY:
Chronic low back pain (CLBP) is a prevalent condition causing significant pain, disability, and reduced quality of life. While various treatments like exercise, NSAIDs, and spinal manipulation are recommended, their effectiveness is limited. Epidural steroid injections can provide short-term relief but may not be cost-effective and have associated risks.

Dexmedetomidine (DXM) is a selective α2-adrenergic agonist with analgesic properties. It has been used as an adjuvant to anesthetics and analgesics to enhance pain relief and reduce opioid consumption. Using DXM in conjunction with local anesthetics for regional blocks has shown promising results in improving analgesia and functional outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had Chronic Lower Back pain defined as persistent pain for more than 6 weeks with manifest affection of daily activities;
* Patients who had Chronic Lower Back pain defined as persistent pain for more than 6 weeks with manifest affection of quality of walking and life;
* Patients who had Chronic Lower Back pain defined as persistent pain for more than 6 weeks maintained on systemic analgesics;
* Patients who were free of exclusion criteria were enrolled in the study.

Exclusion Criteria:

* The presence of osteolytic vertebral lesions;
* The Presence of previous surgical intervention;
* The presence of allergy to the studied drugs;
* Patients of ASA grade >II.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reporting at least a 50% reduction in pain (measured by Numerical Rating Scale) in post-Operative Follow up for Spine Surgery. | 3 months
  Value of Dexmedetomidine injection in Pain Reduction post operatively manifested by recurrence of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia University, Shibīn al Kawm, El Menoufia, Egypt